CLINICAL TRIAL: NCT05732493
Title: Short-course Radiotherapy Combined With CAPOX and Pd-1 Inhibitor for Locally Advanced Colon Cancer: a Randomized, Prospective, Multicentre, Phase II Trial (TORCH-C)
Brief Title: Short-course Radiotherapy Combined With Chemotherapy and Pd-1 Inhibitor for Locally Advanced Colon Cancer(TORCH-C)
Acronym: TORCH-C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoCRT-COLON
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Colon Cancer
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short-course radiotherapy and immunotherapy (Experimental): A total of 60 patients will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody, finally receive the surgery.
  Interventions: Drug: Serplulimab; Radiation: short-term radiotherapy; Drug: Oxaliplatin; Drug: Capecitabine
- chemotherapy (Active Comparator): A total of 60 patients will receive 4 cycles of CAPOX chemotherapy ,then receive the surgery.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Serplulimab — Serplulimab 300mg, d1, q3w
  Arms: short-course radiotherapy and immunotherapy
Radiation: short-term radiotherapy — radiation: 25Gy/5Fx
  Other Names: Shor-course radiotherapy: 25Gy/5Fx
  Arms: short-course radiotherapy and immunotherapy
Drug: Oxaliplatin — 130mg/m2 d1 q3w
Drug: Capecitabine — 1000mg/m2 d1-14 q3w
  Other Names: Xeloda

SUMMARY:
The study evaluates the combination of immunotherapy of PD-1 antibody and chemotherapy and neoadjuvant short-course radiotherapy in locally advanced colon cancer (LACC). Patients are randomly assigned into two prospective groups: treatment group and observerment group. In treatment group, a total of 60 patients will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of capecitabine plus oxaliplatin (CAPOX) chemotherapy and PD-1 antibody, finally receive the surgery. In observerment group: a total of 60 patients will receive 4 cycles of CAPOX chemotherapy, then receive the surgery. The rate of pathologic complete response （pCR）, long-term prognosis and adverse effects will be analyzed.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled, multicenter phase II study, with a design of superior efficacy，to compare the efficacy of neoadjuvant short-course radiotherapy combined with CapOX chemotherapy and PD-1 immunotherapy in locally advanced colon cancer. We will consecutively enrolled patients who were diagnosed with locally advanced colon cancer with T4 stage or bulky nodes. A total of 120 patients will be Randomized 1:1 to the treatment group and observerment group. In observerment group, patients will receive 4 cycles of CAPOX (Capecitabine: 1000mg/m2 d1-14 q3w; Oxaliplatin: 130mg/m2 d1 q3w)chemotherapy, then receive the surgery, followed by 4 cycles of CAPOX. In treatment group, patients will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOXand PD-1 antibody(Serplulimab,300mg d1 q3w), then receive the surgery,followed by 4 cycles of CAPOX.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed adenocarcinoma
2. clinical stage T4 and/or bulky nodes
3. the distance from anal verge more than 15 cm
4. without distance metastases
5. age >=18 years old, female and male
6. KPS >=70
7. without previous anti-cancer therapy or immunotherapy
8. with good compliance
9. signed the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. history of other malignancies within 5 years
3. serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
4. immunodeficiency disease or long-term using of immunosuppressive agents
5. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
6. allergic to any component of the therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | The pCR rate will be evaluated after surgery, an average of 4 weeks
  pCR was defined as the absence, from surgical samples, of malignant cells in the primary site and regional lymph nodes

SECONDARY OUTCOMES:
R0 resection rate | The R0 resection rate will be evaluated after surgery, an average of 4 weeks
  R0 resection refers to the complete removal of the tumor in the operation with microscopically negative margins
3 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 3 years
  Rate of 3 years overall survival
3 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Rate of 3 years disease free survival
Grade 3-4 adverse effects rate | From date of randomization until the date of death from any cause, assessed up to 5 years
  Rate of chemotherapy, radiotherapy and immunotherapy related severe adverse events
3 year local recurrence free survival rate | From date of randomization until the date of first documented local-regional failure, assessed up to 3 years
  Rate of 3 years local recurrence free survival
Surgical complications | The surgery was scheduled 2-4 weeks after the end of neoadjuvant therapy. And the surgical complications were assessed up to 5 years from the surgery
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Li Y, Xia F, Sun Y, Shen L, Wan J, Chen Y, Wang Y, Zhou M, Wu R, Zhou S, Wang Y, Liu F, Cai S, Zhang Z. Study protocol of short-course radiotherapy combined with CAPOX and PD-1 inhibitor for locally advanced colon cancer: a randomised, prospective, multicentre, phase II trial (TORCH-C). BMJ Open. 2024 Feb 2;14(2):e079442. doi: 10.1136/bmjopen-2023-079442. PMID 38309748